CLINICAL TRIAL: NCT05889234
Title: Multimodal Magnetic Resonance Imaging-based Study of Electroconvulsive Efficacy Prediction in Adolescents With Depression: a Multicenter Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: The Second Affiliated Hospital of Chongqing Medical University (Other); Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Xinyu Zhou, Professor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 1stChongqingMUZXY
Record Dates: First submitted 2023-05-26; First posted 2023-06-05 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Major Depressive Disorder; Magnetic Resonance Imaging; Electroconvulsive Therapy
Keywords: adolescent MDD; MECT; Multimodal MRI
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Modified electroconvulsive therapy group: The adolescent MDD receiving modified electroconvulsive therapy and conventional medication.
  Interventions: Device: Modified Electroconvulsive Therapy; Drug: Conventional pharmacotherapy
- Non-modified electroconvulsive therapy group: The adolescent MDD receiving only conventional medication.
  Interventions: Drug: Conventional pharmacotherapy
- Healthy controls group: Healthy adolescents.

INTERVENTIONS:
Device: Modified Electroconvulsive Therapy — MECT is performed using the Thymatron System IV (Somatics LLC, LakeBluff, IL, USA) electroconvulsive therapy (ECT) machine. Prior to ECT, all patients undergo laboratory tests such as routine blood, liver, kidney and thyroid function and an ECG and remain fasted for 12 hours. Initial treatment power is considered by age: percentage of power = age x 0.7. Stimulation power is adjusted according to seizure duration. If the seizure duration is less than 25 seconds, the energy is increased by 5% in the subsequent treatments. Anaesthesia and muscle relaxation were administered with propofol (1.5-2 mg/kg) and succinylcholine (0.5-1 mg/kg), respectively, and subjects were awakened after ECT treatment and adverse effects, such as subjective memory impairment, headache or nausea/vomiting, were recorded. Frequency of ECT treatment: 3-4 times per week for a total of 6-8 sessions
  Groups: Modified electroconvulsive therapy group
Drug: Conventional pharmacotherapy — Conventional pharmacotherapy: SSRIs including fluoxetine, paroxetine, sertraline, cetinopram, fluvoxamine, vortioxetine, escitalopram; SNRIs including venlafaxine, duloxetine; NaSSA including mirtazapine; other antidepressants including trazodone, bupropion, agomelatine; potentiators including aripiprazole, olanzapine, quetiapine, risperidone.
  Groups: Modified electroconvulsive therapy group; Non-modified electroconvulsive therapy group

SUMMARY:
The aim of this project is to investigate the multimodal magnetic resonance brain imaging changes in adolescents with major depressive disorder (MDD) before and after electroconvulsive therapy. Development of a predictive model for the efficacy of electroconvulsive therapy in adolescent MDD.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational study. We will divide the adolescent MDD patients into two groups according to the treatment modality as follows: Group 1 (Modified Electroconvulsive Therapy (MECT), n=60); Group 2 (Non-Modified Electroconvulsive Therapy (Non-MECT), n=60). Patients in group 1 will be treated with MECT according to standard clinical care. Group 2 will receive conventional drug therapy. A healthy control group (n=60) will also be recruited.

The most modern MRI sequences examining brain structure and function are used at 4 time points: at baseline (just before MECT series), the second examination (just after MECT series) and the third and forth (follow-up) examination (3 and 6 months after MECT series). Blood, urine and feces samples and the evaluation of clinical effect and side-effects to MECT are performed at the same time points.

The primary outcome for the treatment phase is the treatment remission rate and response rate. The secondary outcomes included: symptom scale, Quality of life, Sleep therapy, Symptoms of anxiety, Rumination and safety assessment.

ELIGIBILITY:
Inclusion criteria for the modified electroconvulsive therapy (MECT) and non-modified electroconvulsive therapy (Non-MECT) groups:

1. Age 13-18 years.
2. Meeting a diagnosis of depression (MDD) from the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) based the Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL).
3. A score of ≥40 on the Childhood Depression Rating Scale-Revised (CDRS-R).
4. Adequate audiovisual level to be able to complete this study.
5. Signed informed consent and signed by the subject and guardian.

Healthy control group inclusion criteria.

1. Age 13-18 years.
2. Sufficient audio-visual level to be able to complete the study.
3. Signed informed consent form and signed by the subject and guardian.

Exclusion criteria for the modified electroconvulsive therapy (MECT) and non-modified electroconvulsive therapy (Non-MECT) groups:

1. The presence or previous presence of a serious medical, neurological or psychiatric condition (except in patients with MDD; anxiety co-morbidity is not considered an exclusion criterion, provided that MDD is the primary diagnosis and the main reason for seeking life-saving treatment).
2. Patients who have received electroconvulsive therapy within the last 12 months.
3. Patients with a history of substance, drug abuse.
4. Contraindications to anaesthesia or MRI.
5. Lactating women or pregnant women.
6. Left-handedness.

Exclusion criteria for healthy controls:

1. Presence or previous serious medical, neurological or psychiatric illness.
2. Patients with a history of substance or drug abuse.
3. Contraindications to MRI.
4. Lactating women or pregnant women.
5. Left-handedness.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients accepted for ECT or medication treatment in the inpatient adolescent MDD patients. According to treatment modality in two groups, as follows: Group 1 (modified electroconvulsive therapy (MECT) ,n=60); Group 2 (Non-modified electroconvulsive therapy(Non-MECT), n=60). Each enrolled participant in group 1 will undergo an index course of MECT, following standard clinical care. Group 2 will receive conventional drug therapy. At the same time, a healthy control group (n=60) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-11-06 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in CDRS-R (Children's Depression Rating Scale, Revised) scores | The treatment period was baseline, 2-4 weeks. The follow-up period was 1 month, 3 months, 6 months.
  Clinical response (≥ 50% reduction in CDRS-R scores from baseline).

SECONDARY OUTCOMES:
Changes in BDI (Beck's Depression Inventory) scores | The treatment period was baseline, 2-4 weeks. The follow-up period was 1 month, 3 months, 6 months.
  The severity of depression symptom.
Changes in SCARED (Screen for Child Anxiety Related Disorders) scores | Baseline of treatment period, 2-4 weeks; The follow-up period was 3 months, 6 months
  The severity of Anxiety symptom.
Changes in suicide risk on C-SSRS (Columbia Suicide Severity Rating Scale) scores | Baseline of treatment period, 2-4 weeks; The follow-up period was 3 months, 6 months
  The severity of the suicide risk.
Changes in PSQI (Pittsburgh Sleep Quality Index) scores | Baseline of treatment period, 2-4 weeks; The follow-up period was 3 months, 6 months
  Measures of sleep status.
Changes in PedsQL4.0 (The Pediatric Quality of Life Inventory 4.0) scores | Baseline of treatment period, 2-4 weeks; The follow-up period was 3 months, 6 months
  Measures of children's quality of life.
Changes in CGI-S (Clinical Global Impressions-Severity Scales) scores | Baseline of treatment period, 2-4 weeks
  Measures of clinical impression severity.
Changes in CGI-I (Clinical Global Impressions-Improvement Scales) scores | The treatment period was 2-4 weeks
  Measures of clinical general Impression scale.
Changes in RSS (Ruminative Responses Scale) scores | Baseline of treatment period, 2-4 weeks; The follow-up period was 3 months, 6 months
  Measures of negative thinking.
Assessment of CTQ（Childhood Trauma Questionnaire） | Baseline of treatment period
  Measures of childhood trauma.
Assessment of OB/VQ（Olweus Bully/Victim Questionnaire） | Baseline of treatment period
  Measures of bully/victim problems.
Changes in AE（Adverse Event）Scale | The treatment period was 2-4 weeks; The follow-up period was 1 month, 3 months, 6 months.
  Measures of any untoward medical orrurrence in a patient or clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.
Assessment of SAE（Serious Adverse Event）Scale | The treatment period was 2-4 weeks; The follow-up period was 1 month, 3 months, 6 months.
  Measures of adverse medical events.
Changes in THINC-it | Baseline of treatment period, 2-4 weeks; The follow-up period was 3 months, 6 months
  Measures of cognition function.
Changes in functional MRI | Baseline of treatment period, 2-4 weeks; The follow-up period was 3 months, 6 months
  Resting state MRI, measurement of functional connectivity.
Changes in structural MRI T1 and T2 | Baseline of treatment period, 2-4 weeks; The follow-up period was 3 months, 6 months
  Measures of brain structure.
Changes in Cerebral Blood Flow | Baseline of treatment period, 2-4 weeks; The follow-up period was 3 months, 6 months
  Estimated by Arterial Spin Labeling MRI.
Changes in concentration of Glu and GABA in ACC | Baseline of treatment period, 2-4 weeks; The follow-up period was 3 months, 6 months
  MR Spectroscopy og the ACC, measures of neuronal integrity.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Province, China